CLINICAL TRIAL: NCT07398209
Title: Combining 4D MRI and 4DCT for Personalized Volumetric Motion Monitoring in Lung Radiation Therapy
Brief Title: GCC 2546- Motion Management
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Amit Sawant, Principal Investigator, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HP-00114565
Record Dates: First submitted 2026-02-02; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Lung Cancer (NSCLC); Radiation
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Imaging (Experimental): At baseline, patients will receive a 4D CT Simulation (standard of care) along with a 4D MRI with surface monitoring (research).
  During their radiation treatment, they will receive additional fluoroscopy imaging and surface monitoring.
  Interventions: Other: MRI

INTERVENTIONS:
Other: MRI — Baseline 4D CT Simulation and 4S MRI with surface monitoring through EndoScout vest, followed by fluoroscopy and additional surface monitoring while undergoing daily radiation.
  Other Names: Fluoroscopy; Surface Monitoring

SUMMARY:
The purpose of this study is to assess a real time motion tracking of lung tumors and important organs next to the tumor while breathing during a participant's radiation treatment. This will be assessed through a four-dimensional magnetic resonance imaging (MRI) scan before starting your radiation treatment and x-ray fluoroscopy images that are taken during radiation

ELIGIBILITY:
Inclusion Criteria:

1. Adult (≥18 years) patients (both sexes) with histologically diagnosed Stage II-IIIb NSCLC
2. Patients to be treated with definitive external beam photon radiotherapy with or without systemic therapy (e.g., chemotherapy, immunotherapy).
3. No restrictions on number radiotherapy fractions, or location/number of lesions
4. ECOG performance status ≤ 3
5. Ability to undergo MRI scans
6. Patient has signed informed consent document and agreed to study procedures

Exclusion Criteria:

1. Pre-existing contraindications for MRI, such as any MRI-conditional or MRI-unsafe foreign objects within the body, non-removable ear cochlear or eye implant, aneurysm clip, cardiac pacemaker/wires, internal defibrillator, tissue expander, recent stent placement, penile prosthesis, medication patch, artificial limb, pregnancy, and claustrophobia
2. Women who are pregnant or trying to get pregnant (self-reported)
3. Pain in supine position or inability to raise arm above head in supine position

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2028-04 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
To investigate if time-resolved, multicycle volumetric motion modeling and monitoring gives improved spatiotemporal localization of the tumor target and OARs compared to current standard-of-care 4DCT-based motion modeling and monitoring | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Amit Sawant, PhD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland Greenebaum Cancer Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No